CLINICAL TRIAL: NCT02189902
Title: Botswana Vitamin D Supplementation Study in HIV/AIDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Principal Investigator, Virginia Stallings, Professor of Pediatrics, Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812323
Record Dates: First submitted 2014-07-11; First posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-07

CONDITIONS: HIV
Keywords: Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4000 IU/d of D3 by mouth for 12 weeks (Active Comparator): 4000 IU/d of D3 by mouth for 12 weeks
  Interventions: Dietary Supplement: 4000 IU/d D3 over 12 weeks
- 7000IU/d of D3 by mouth for 12 weeks (Experimental): 7000IU/d of D3 by mouth for 12 weeks
  Interventions: Dietary Supplement: 7000 IU/d D3 over 12 weeks

INTERVENTIONS:
Dietary Supplement: 4000 IU/d D3 over 12 weeks
  Arms: 4000 IU/d of D3 by mouth for 12 weeks
Dietary Supplement: 7000 IU/d D3 over 12 weeks
  Arms: 7000IU/d of D3 by mouth for 12 weeks

SUMMARY:
The goal is to determine the vit D supplementation dose that safely results in optimal serum vitamin D (25D) concentrations in HIV-infected children and adults living in Botswana. To do this the investigators will test two oral daily doses (4000 vs. 7000 IU) of cholecalciferol (D3) dietary supplement over a 12-week period in 60 children and adults with HIV/AIDS living in Botswana (5.0 to 50.9 yrs), to assess safety as determined by serum calcium and 25D concentrations and efficacy to replete vit D status as determined by achieving a minimum serum 25D concentration of 32 ng/mL (80 nmol/L).

DETAILED DESCRIPTION:
Many people living with HIV/AIDS in African countries are vit D deficient or insufficient. Vit D deficiency in HIV/AIDS may be due to low dietary vit D intake, increased requirements, malabsorption, specific drug therapies (antiretrovirals, in particular), reduced outdoor physical activity, reduced vit D synthesis from UV light exposure in dark skin pigmented individuals, or unknown HIV-associated factors. Vit D deficiency likely contributes to abnormal immune status and increased inflammatory state, and to poor growth, bone, and muscle function, and may contribute to risk for tuberculosis (TB) infection. The goal is to determine the vit D supplementation dose that safely results in optimal serum 25D concentrations in HIV-infected children and adults living in Botswana.

To do this the investigators will test two oral daily doses (4000 vs. 7000 IU) of cholecalciferol (D3) dietary supplement over a 12-week period in 60 children and adults with HIV/AIDS living in Botswana (5.0 to 50.9 yrs), to assess safety as determined by serum calcium and 25D concentrations and efficacy to replete vit D status as determined by achieving a minimum serum 25D concentration of 32 ng/mL (80 nmol/L).

ELIGIBILITY:
Inclusion Criteria:

* HIV infection
* Ages 5.0 to 50.9 y
* In usual state of good health
* Subject and/or family commitment to the 12-week study

Exclusion Criteria:

* Other chronic health conditions unrelated to HIV/AIDS that may affect nutritional status
* Use of vit D supplementation above 400 IU/d

Ages: 5 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2012-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To test the efficacy of two oral doses (4000 vs 7000 IU/d) of cholecalciferol (D3) in 60 children and adults (5.0 to 50.9 y) with HIV/AIDS to replete vit D status (achieving a minimum serum 25D concentration of 32 ng/mL). | 12 weeks
  To test two oral doses (4000 vs 7000 IU/d) of cholecalciferol (D3) over a 12-week period in 60 children and adults (5.0 to 50.9 y) with HIV/AIDS to assess 25D concentrations and efficacy to replete vit D status as determined by achieving a minimum serum 25D concentration of 32 ng/mL.
To test the safety of two oral doses (4000 vs 7000 IU/d) of cholecalciferol (D3) over a 12-week period in 60 children and adults (5.0 to 50.9 y) with HIV/AIDS as determined by serum calcium. | 12 weeks
  To test two oral doses (4000 vs 7000 IU/d) of cholecalciferol (D3) over a 12-week period in 60 children and adults (5.0 to 50.9 y) with HIV/AIDS to assess safety as determined by serum calcium.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Stallings, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Princess Marina Hospital, Gaborone, Botswana

REFERENCES:
- [Derived] Steenhoff AP, Schall JI, Samuel J, Seme B, Marape M, Ratshaa B, Goercke I, Tolle M, Nnyepi MS, Mazhani L, Zemel BS, Rutstein RM, Stallings VA. Vitamin D(3)supplementation in Batswana children and adults with HIV: a pilot double blind randomized controlled trial. PLoS One. 2015 Feb 23;10(2):e0117123. doi: 10.1371/journal.pone.0117123. eCollection 2015. PMID 25706751